CLINICAL TRIAL: NCT00003765
Title: A Trial of 06-BG and BCNU in Children With CNS Tumors
Brief Title: O6-benzylguanine and Carmustine in Treating Children With Refractory CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01842; POG-9870; CDR0000066891 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2007-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood craniopharyngioma; childhood central nervous system germ cell tumor; childhood oligodendroglioma; childhood choroid plexus tumor; recurrent childhood brain stem glioma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood visual pathway glioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Choroid Plexus Neoplasms; Optic Nerve Glioma; Astrocytoma; Medulloblastoma; Familial ependymoma | interventions — O(6)-benzylguanine; Carmustine

ARMS (1):
- Arm I (Experimental): Patients receive O6-benzylguanine IV over 1 hour, then, 1 hour later, carmustine IV is administered over 1 hour. Treatment is repeated every 6 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients each receive escalating doses of carmustine until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose level at which fewer than 2 of 6 patients experience dose limiting toxicity (DLT). If myelosuppression is the DLT, stratum 1 is closed and patients are accrued to stratum 2. If neutropenia is the DLT in stratum 2, patients receive filgrastim (G-CSF) subcutaneously beginning on day 2 and continuing until blood counts recover.
  Interventions: Drug: O6-benzylguanine; Drug: carmustine

INTERVENTIONS:
Drug: O6-benzylguanine
Drug: carmustine

SUMMARY:
Phase I trial to study the effectiveness of O6-benzylguanine and carmustine in treating children who have refractory CNS tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and the dose limiting toxicity of carmustine administered after O6-benzylguanine in children with refractory primary CNS tumors.

II. Determine a safe and tolerable dose of carmustine administered after O6-benzylguanine to be used in phase II studies.

III. Determine the pharmacokinetics of O6-benzylguanine and its metabolite, O6-benzyl-8-oxoguanine, in these patients.

IV. Seek preliminary evidence of antitumor activity of this regimen in these patients.

V. Evaluate the acute and chronic toxicities, and describe cumulative toxicity, in patients treated with multiple courses of this regimen.

OUTLINE: This is a dose escalation study of carmustine.

Patients receive O6-benzylguanine IV over 1 hour, then, 1 hour later, carmustine IV is administered over 1 hour. Treatment is repeated every 6 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients each receive escalating doses of carmustine until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose level at which fewer than 2 of 6 patients experience dose limiting toxicity (DLT). If myelosuppression is the DLT, stratum 1 is closed and patients are accrued to stratum 2. If neutropenia is the DLT in stratum 2, patients receive filgrastim (G-CSF) subcutaneously beginning on day 2 and continuing until blood counts recover. Patients are followed every 6 months for 4 years, then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven CNS tumor that is refractory to conventional therapy or for which no effective therapy is known
* Histological requirement may be waived for brainstem and optic gliomas
* Stratum 2: No bone marrow involvement

PATIENT CHARACTERISTICS:

* Age: 21 and under
* Performance status: Karnofsky 50-100% OR Lansky 50-100%
* Life expectancy: At least 8 weeks
* Absolute neutrophil count at least 1500/mm3
* Platelet count at least 100,000/mm3 (stratum 2: at least 125,000/mm3)
* Hemoglobin at least 8 g/dL
* Bilirubin less than 1.5 mg/dL
* SGOT/SGPT no greater than 2.5 times normal
* Creatinine or GFR normal for age
* If required, DLCO must be 80% of normal and patient old enough to cooperate for DLCO test
* Neurologic deficits must be stable for at least 2 weeks prior to study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study

PRIOR CONCURRENT THERAPY:

* At least 7 days since prior biologic therapy or immunotherapy and recovered
* At least 6 months since prior bone marrow transplant (stratum 1 only)
* At least 7 days since prior growth factors
* No concurrent filgrastim (G-CSF) prophylaxis
* Stratum 2: No prior bone marrow transplantation
* At least 2 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea) and recovered
* Stratum 2: No greater than 2 prior chemotherapy regimens
* No prior nitrosourea therapy
* If receiving dexamethasone, must be on stable or decreasing dose for at least 2 weeks prior to study
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months since prior substantial bone marrow radiation, total body irradiation, hemipelvic radiotherapy, or total abdominal/pelvic/chest or mantle/Y ports radiotherapy
* Recovered from prior radiotherapy
* Stratum 2: No prior central axis radiation
* No other concurrent anticancer or investigational agents

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 1999-05; Primary Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Adams, MD, Study Chair — University of Vermont
Locations (56):
- United States (51):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - City of Hope National Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center, Gainesville, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Graham Children's Health Center, Asheville, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (3):
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Adams DM, Zhou T, Berg SL, Bernstein M, Neville K, Blaney SM; Children's Oncology Group. Phase 1 trial of O6-benzylguanine and BCNU in children with CNS tumors: a Children's Oncology Group study. Pediatr Blood Cancer. 2008 Mar;50(3):549-53. doi: 10.1002/pbc.21362. PMID 17941066